CLINICAL TRIAL: NCT03402126
Title: Tachy Prediction Download Study
Acronym: TPD
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: TPD Study
Record Dates: First submitted 2017-12-18; First posted 2018-01-18 (Actual); Results first posted 2021-11-16 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Ventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- TPD RAMWare Download: Subjects who qualify and consent to participate in the TPD study will have TPD RAMWare injected into their device to collect data.
  Interventions: Other: TPD RAMWare

INTERVENTIONS:
Other: TPD RAMWare — TPD RAMWare injected into enrolled subject's Implantable cardioverter-defibrillator (ICD) device for use

SUMMARY:
The purpose of the Medtronic Tachy Prediction Download (TPD) study is to collect data from an implantable cardiac defibrillator (ICD) device that will be used to identify markers for imminent onset of ventricular arrhythmias.

DETAILED DESCRIPTION:
The TPD Study is a prospective, non-randomized, non-interventional, multi-site data collection clinical study to collect ICD longitudinal data that may be used to develop a VT/VF prediction algorithm. The study subjects will include patients currently implanted, or who will be implanted with a market-approved Medtronic Evera MRI® ICD.

ELIGIBILITY:
Inclusion Criteria:

* Subject is implanted or will be implanted, with an Evera MRI device with properly functioning Medtronic tachycardia lead placed in the right ventricle (with or without atrial lead) with remaining device longevity of 4 years or more for:

  * Secondary Prevention or,
  * Primary Prevention and has had a device treated VT/VF or a device recorded episode of sustained VT/VF
* Subject is ≥ 18 years old
* Subject has previously documented history of VT/VF
* Subject must be willing and able to use Medtronic CareLink network monitoring system
* Subject provides signed and dated authorization and/or consent per institution and local requirements
* Subject is willing and able to comply with the protocol

Exclusion Criteria:

* Subject who received device for Primary Prevention indication and who has not had either a device treated VT/VF episode or a device recorded episode of sustained VT/VF
* Subject is enrolled in a concurrent study that may confound the results of this study, without documented pre-approval from a Medtronic study manager
* Subject has chronic AF
* Subject has inherited disorders of ion transport mechanisms that predispose the subject to sudden death ("Channelopathies"): Long QT and Brugada Syndromes
* Subject with multiple implanted active devices that may cause an interruption of a transmission of device data to CareLink
* Subject has active electronic medical device other than an ICD
* Subject requires more than 25% atrial or ventricular pacing
* Subject has medical conditions that would limit study participation (per investigator judgment)
* Subject has projected life expectancy of less than 1 year
* Subject is pregnant or plans to be pregnant over the next year (females of child-bearing potential must have a negative pregnancy test within one week of enrollment and must practice a reliable form of birth control while enrolled in the study)
* Subject meets exclusion criteria required by local law (e.g. age, breastfeeding, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study subjects will include patients currently implanted, or who will be implanted with a market-approved Medtronic Evera MRI® ICD.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Brown, Study Director — Medtronic
Locations (16):
- United States (15):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Iowa Heart Center, Des Moines, Iowa
  - Beaumont Hospital - Royal Oak, Royal Oak, Michigan
  - CentraCare Heart & Vascular Center, Saint Cloud, Minnesota
  - United Heart and Vascular Clinic, Saint Paul, Minnesota
  - Saint Lukes Hospital of Kansas City, Kansas City, Missouri
  - Bryan Heart, Lincoln, Nebraska
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Carolinas Medical Center, Charlotte, North Carolina
  - Cape Fear Heart Associates, Wilmington, North Carolina
  - Mount Carmel East, Columbus, Ohio
  - Oklahoma Heart Hospital Research Foundation, Oklahoma City, Oklahoma
  - The Stern Cardiovascular Foundation, Germantown, Tennessee
  - Centennial Heart Cardiovascular Consultants, Nashville, Tennessee
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
- Princess Margaret Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- TPD RAMWare Download: Subjects who qualify and consent to participate in the TPD study will have TPD RAMWare injected into their device to collect data.
  TPD RAMWare: TPD RAMWare injected into enrolled subject's device.
Period: Overall Study
Arm/Group | TPD RAMWare Download
Started | 138
Completed | 76
Not Completed | 62
Not completed — Lost to Follow-up | 6
Not completed — Protocol Violation | 10
Not completed — Sponsor request/Study termination | 29
Not completed — Study product no longer in use | 1
Not completed — Technical problems | 1
Not completed — Withdrawal by Subject | 6
Not completed — Physician Decision | 2
Not completed — upgrade to Cardiac Resynchronization Therapy-Defibrillator/stage IV cancer | 3
Not completed — Death | 4

BASELINE CHARACTERISTICS:
Population: Total number of all participants for whom baseline characteristics were measured and received the Ramware injection. 138 participants were assessed for eligibility but only 128 had baseline characteristics measured and received the Ramware injected. 10 participants did not receive Ramware injection and undergo baseline characteristic measurements due to 8 experiencing screen failures, 1 experiencing noncompliance, and 1 being removed due to physician decision.
Groups:
- TPD RAMWare Injected: Subjects who qualify and consent to participate in the TPD study will have TPD RAMWare injected into their device to collect data.
  TPD RAMWare: TPD RAMWare injected into enrolled subject's device.
Arm/Group | TPD RAMWare Injected
Number analyzed (Participants) | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 104
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 126
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 29
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 81
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  Hong Kong | 28
  United States | 100
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.8 (6.9)
Weight [Mean (Standard Deviation); unit: kg] | 90.1 (22.5)
Height [Mean (Standard Deviation); unit: cm] | 173.8 (10.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Device Detected Ventricular Tachycardia/Ventricular Fibrillation Episodes
Description: This was a data collection study collecting data when implanted device detected Ventricular Tachycardia/Ventricular Fibrillation.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | TPD RAMWare Download
Number analyzed (Participants) | 128
Participants
  Participants with device detected ventricular tachycardia/ventricular fibrillation episodes | 31
  Participants with no device detected ventricular tachycardia/ventricular fibrillation episode | 97

ADVERSE EVENTS:
Time Frame: 1 year (12 months)
Arm/Group | TPD RAMWare Download
All-Cause Mortality (participants affected / at risk) | 4/128
Serious Adverse Events (participants affected / at risk) | 0/128
Other Adverse Events (participants affected / at risk) | 0/128

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Participating Institution and PI agree that it will not independently publish, publicly disclose, present or discuss any results of or information pertaining to the Study until a multi-center publication is released; provided however, that if a multicenter publication is not released within one year after completion of the Study at all Study sites, Participating Institution and PI will have the right to publish the results of and information pertaining to their activities.

DOCUMENTS (2):
  • Study Protocol (2017-08-01): https://cdn.clinicaltrials.gov/large-docs/26/NCT03402126/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-21): https://cdn.clinicaltrials.gov/large-docs/26/NCT03402126/SAP_001.pdf